CLINICAL TRIAL: NCT00656682
Title: Primary Care Community Partnerships to Prevent Diabetes
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ronald Ackermann, Senior Associate Dean for Public Health Director, Institute for Public Health and Medicine, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R18DK079855 (NIH); R18DK079855 (NIH)
Record Dates: First submitted 2008-04-10; First posted 2008-04-11 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2014-08

CONDITIONS: Hyperglycemia; Obesity; Diabetes Mellitus
Keywords: Prevention & Control; Hyperglycemia; Obesity; Diabetes Mellitus; Cost Benefit Analysis
MeSH Terms: conditions — Hyperglycemia; Obesity; Diabetes Mellitus | interventions — Nutritionists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietitian Counseling Alone (Active Comparator): Primary care-based identification of pre-diabetes with brief counseling by a dedicated registered dietitian. Registered Dietitian Counseling Alone
  Interventions: Behavioral: Dietitian Counseling Alone
- Dietitian Plus Community Group Lifestyle (Experimental): Primary care-based identification of pre-diabetes with brief counseling by a dedicated registered dietitian, PLUS free-of-charge access to a group-based diabetes prevention lifestyle intervention offered by the community. Dietitian Counseling Plus Community Group Lifestyle Intervention.
  Interventions: Behavioral: Dietitian Plus Community Group Lifestyle

INTERVENTIONS:
Behavioral: Dietitian Counseling Alone — Primary care-based identification of pre-diabetes with brief counseling by a dedicated registered dietitian
  Arms: Dietitian Counseling Alone
Behavioral: Dietitian Plus Community Group Lifestyle — Primary care-based identification of pre-diabetes with brief counseling by a dedicated registered dietitian, PLUS free-of-charge access to a group-based lifestyle intervention offered by the Community to prevent diabetes
  Arms: Dietitian Plus Community Group Lifestyle

SUMMARY:
The purpose of this study is to determine if providing free-of-charge access to a group-based lifestyle intervention delivered in partnership with the community is cost-effective for the prevention of type 2 diabetes.

DETAILED DESCRIPTION:
Randomized controlled trials have shown that modest lifestyle changes can prevent or delay the onset of diabetes in adults with pre-diabetes. Unfortunately, despite the increasing prevalence of pre-diabetes and diabetes in all facets of the population, intervention programs needed to achieve these goals are costly and remain unavailable in most clinical settings. Over the past 3 years, we have demonstrated the feasibility of training community instructors to deliver a group-based adaptation of the Diabetes Prevention Program (DPP) lifestyle intervention. In this pilot research, this new delivery model achieves a level of weight reduction that was associated with diabetes prevention and improved cardiometabolic risk factor control in the DPP. This new, large-scale randomized effectiveness trial is designed to evaluate the costs and effectiveness of a partnered approach to identify adults with pre-diabetes in primary care settings, deliver brief advice for diabetes prevention, and provide access to a group-based adaptation of the DPP lifestyle intervention offered by the community. This study will compare costs and outcomes to a standard care, brief clinical counseling approach delivered by Registered Dietitians.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Body-mass index of 24 kg/m2 or greater
* Fasting Blood Glucose 100 - 125 mg/dl, OR 2-hour Post-challenge Capillary Glucose 140 - 199 mg/dl

Exclusion Criteria:

* Cancer requiring treatment in the past 5 years
* Uncontrolled hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg
* Heart attack, stroke, or transient ischemic attack in the past 6 months,
* Chronic obstructive airways disease or asthma requiring home oxygen
* Other chronic disease or condition, such as advanced arthritis, that could limit ability to become physically active or limit life span to <5 years
* Pregnancy
* Existing diagnosis of diabetes mellitus
* Fasting capillary blood glucose > 125 mg/dl
* 2-hour post-challenge capillary blood glucose > 199 mg/dl
* History of anti-diabetic medication use (oral agents or insulin) except during gestational diabetes
* Self-report of a medication known to lead to hyperglycemia (oral steroids, antipsychotics, anti-epileptics)
* Self-report of disease associated with disordered glucose metabolism: Cushing's syndrome; acromegaly; pheochromocytoma; chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2008-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
% Change in Body Weight | 12 months
  (weight in kg at 12 months - weight in kg at baseline) / (weight in kg at baseline)

SECONDARY OUTCOMES:
% Change in Blood Total Cholesterol | 12 months
  (total blood cholesterol concentration at 12 months - total blood cholesterol concentration at baseline) / (total blood cholesterol concentration at baseline)
% Change in glycosylated hemoglobin | 12 months
  (HbA1c % at 12 months - HbA1c % at baseline) / (HbA1c % at baseline)
% Change in Blood Pressures | 12 months
  (mean SBP at 12 months - mean SBP at baseline) / (mean SBP at baseline); (mean DBP at 12 months - mean DBP at baseline) / (mean DBP at baseline)
Changes in Dietary Composition | 12 months
  NHIS Multifactor Screener: Change in % dietary kcal from fat at 12 months (est % dietary Kcal from fat at 12 months - est % dietary Kcal from fat at baseline)
Changes in Physical Activity | 12 months
  Paffenbarger PAQ: (Total Kcal/week energy expenditure from walking, stairs, and leisure time activity at 12 months - Total Kcal/week energy expenditure from walking, stairs, and leisure time activity at Baseline)
Incremental Costs | 12 months
Incremental Health State Utility | 12 months
% Change in Body Weight | 6 months
  (weight in kg at 6 months - weight in kg at baseline) / (weight in kg at baseline)
% Change in Body Weight | 24 months
  (weight in kg at 24 months - weight in kg at baseline) / (weight in kg at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Ackermann, MD, MPH, Principal Investigator — Northwestern University School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No